CLINICAL TRIAL: NCT06742125
Title: Drug-Coated Balloon Versus Drug-Eluting Stent in Patient With ST-Segment Elevation Myocardial Infarction
Acronym: DCB-STEMI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: The First Affiliated Hospital of Zhengzhou University (Other); Peking University First Hospital (Other); Suzhou Municipal Hospital (Other); First Affiliated Hospital of Ningbo University (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-0936
Record Dates: First submitted 2024-12-09; First posted 2024-12-19 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-05

CONDITIONS: ST-elevation Myocardial Infarction (STEMI)
Keywords: Drug-coated balloon; Drug-eluting stent; ST-elevation myocardial infarction (STEMI)
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Drug-Eluting Stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DCB group (Experimental): STEMI patients undergo revascularization using DCB
  Interventions: Device: Drug-coated balloon (DCB)
- DES group (Active Comparator): STEMI patients undergo revascularization using DES
  Interventions: Device: Drug-eluting stent (DES)

INTERVENTIONS:
Device: Drug-coated balloon (DCB) — Drug-coated balloon treatment of target lesions in patients with STEMI undergoing percutaneous coronary intervention.
  Arms: DCB group
Device: Drug-eluting stent (DES) — Drug-eluting stent treatment of target lesions in patients with STEMI undergoing percutaneous coronary intervention.
  Arms: DES group

SUMMARY:
Acute ST-segment elevation myocardial infarction (STEMI) is a life-threatening emergency requiring immediate intervention. The incidence of premature coronary artery disease (PCAD) is rising rapidly in China; its long-term prognosis remains poor and it frequently progresses to acute myocardial infarction, necessitating high-risk therapies such as primary percutaneous coronary intervention (PCI) or coronary artery bypass grafting, thereby imposing enormous economic and psychological burdens on patients and their families. Moreover, the cumulative 6-year rate of death or myocardial infarction after implantation of the latest-generation drug-eluting stents still reaches 15%, and management of stent failure is extremely challenging. Drug-coated balloon (DCB) angioplasty-representing the "leave-nothing-behind" paradigm-is a highly promising option in young subjects. Accumulating clinical evidence demonstrates that DCB provides favorable efficacy across a broad spectrum of lesions, including small-vessel and large-vessel de novo disease, bifurcation lesions, and in-stent restenosis. Nevertheless, high-quality data on the impact of DCB angioplasty in de novo large-vessel disease and in the setting of acute STEMI are still lacking.

DETAILED DESCRIPTION:
Objectives of Study:

Compare the clinical outcomes of drug-coated balloon (DCB) and drug-eluting stent (DES) treatment in patients with ST-segment elevation myocardial infarction (STEMI).

Design of Study:

Investigator-Initiated，Open Label，Prospective，Multicenter，Randomized Clinical Trial.

Patients Selected： This study aims to STEMI patients who have successfully completed lesion pretreatment in multiple medical centers in China. Patients who meet the inclusion criteria and have no exclusion criteria will be randomly assigned 1:1 to the drug coated balloon group and drug eluting stent group, totaling 1244 cases (622 cases per group).

Primary Endpoints:

Patient-oriented composite endpoints (POCE) within 12 months, including all-cause mortality, any myocardial infarction, any stroke, and any revascularization.

Hypothesis:

The 12-month POCE rate in the DCB group of STEMI patients is not inferior to that of the DES group.

Sample's Size:

Sample size calculation based on the event rates of previous trials. DES group had a predetermined events' rate of 8.0%, the DCB group had a predetermined events' rate of 6.3%.

* Design: Non-inferiority, delta=2.5%
* Ratio of Specimen: DCB : DES= 1:1
* Type I Error (α): Single side 2.5%
* Duration of Participation: 2 years
* Setting: The 12-month clinical events' rates for the DCB group and DES group were 6.3% and 8.0%, respectively.
* Statistical Testing Efficiency (1- β): 80%
* Main Statistical Methods: Kaplan-meier survival analysis using log rank testing
* Dropout Rate: 5% of all the patients Based on the above assumptions and dropout rate, we need to include a total of 1244 cases (622 cases per group).

ELIGIBILITY:
Inclusion Criteria:

1. . Age of Patients ≥18 years old;
2. Acute myocardial infarction patients with onset symptoms<48 hours require emergency PCI;
3. . Diagnosis: Chest pain and other ischemic symptoms accompanied by ST segment elevation in at least two adjacent leads on electrocardiogram (① V2 or V3 lead: male<40 years ≥ 0.25mV, ≥ 40 years ≥ 0.2mV; Female ≥1.5mV；② Other leads ≥ 1mV), or new left bundle branch block occurs;
4. Criminal blood vessels with clear requirements for emergency PCI;
5. Coronary artery in situ lesions, with a visual reference lumen diameter of ≥ 2mm and ≤ 4mm; Lesion's length<40mm；
6. After thrombus aspiration and pre dilation, the lesion stenosis is ≤ 50% and there is no C-type or above dissection.
7. He/she or his/her legal representative voluntarily participates in this study and signs an informed consent form.

Exclusion Criteria:

1. The patient has allergies or contraindications to the following medications: Heparin, Aspirin, Clopidogrel, Prasugrel, Ticagrelor, Cilostazol, Indobufen, Contrast Medias (Patients with clear contrast agent allergies such as rash but can be controlled with effective drugs such as glucocorticoids and diphenhydramine in advance can be selected);
2. The patient has active pathological bleeding;
3. History of significant gastrointestinal or urogenital bleeding or bleeding tendency within 3 months prior to surgery, known coagulation disorders (including heparin induced thrombocytopenia);
4. Patients who are pregnant or have the intention to become pregnant during the period of research;
5. Non cardiogenic combined lesions show an expected life expectancy of less than one year;
6. Left main trunk's stenosis ≥ 50%
7. History of coronary artery bypass grafting in the past;
8. Intubation or mechanical ventilation status;
9. . Cardiogenic Shock
10. . Without signature on informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1244 (Estimated)
Dates: Start 2025-05-31 (Actual); Primary Completion 2032-01-01 (Estimated); Study Completion 2032-01-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of patient-oriented composite endpoints (POCE) (Direct measurement and coronary angiography) | 12 months
  POCE including all-cause mortality, any stroke, any myocardial infarction (MI), and any revascularization, will be obtained through follow-up of subjects.

SECONDARY OUTCOMES:
Incidence of patient-oriented composite endpoints (POCE) (Direct measurement and coronary angiography) | 36 months, 60 months
  POCE including all-cause mortality, any stroke, any myocardial infarction (MI), and any revascularization, will be obtained through follow-up of subjects.
Incidence of target vessel failure (Direct measurement and coronary angiography) | 12 months
  Target vessel failure (a composite of cardiac death, target-vessel MI, or target vessel revascularization) will be obtained through follow-up of subjects.
Incidence of all-cause mortality (Direct measurement) | 36 months, 60 months
  All-cause mortality will be obtained through follow-up of subjects.
Incidence of non-fatal MI (Direct measurement) | 36 months, 60 months
  Non-fatal MI will be obtained through follow-up of subjects.
Incidence of any revascularization (coronary angiography) | 36 months, 60 months
  Any revascularization will be obtained through follow-up of subjects.
Incidence of all-cause and cardiac death (Direct measurement) | 12 months, 36 months, 60 months
  All-cause and cardiac death will be obtained through follow-up of subjects.
Incidence of any non-fatal MI without peri-procedural MI (Direct measurement) | 12 months, 36 months, 60 months
  Any non-fatal MI without peri-procedural MI will be obtained through follow-up of subjects.
Incidence of any non-fatal MI with peri-procedural MI (Direct measurement) | 12 months, 36 months, 60 months
  Any non-fatal MI with peri-procedural MI will be obtained through follow-up of subjects.
Incidence of any target vessel/lesion revascularization (Coronary angiography) | 12 months, 36 months, 60 months
  Any target vessel/lesion revascularization will be obtained through follow-up of subjects.
Incidence of any non-target vessel/lesion revascularization (Coronary angiography) | 12 months, 36 months, 60 months
  Any non-target vessel/lesion revascularization will be obtained through follow-up of subjects.
Incidence of any revascularization (ischemia-driven or all) (Coronary angiography) | 12 months, 36 months, 60 months
  Any revascularization (ischemia-driven or all) will be obtained through follow-up of subjects.
Incidence of non-fatal stroke (ischemic and hemorrhagic) (Direct measurement) | 12 months, 36 months, 60 months
  Non-fatal stroke (ischemic and hemorrhagic) will be obtained through follow-up of subjects.
CRP and POCE | 12 months, 36 months, 60 months
  Prognostic value of CRP on POCE

CONTACTS AND LOCATIONS:
Overall Officials: Jun Jiang, Study Director — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No